CLINICAL TRIAL: NCT01958424
Title: The Influence of Metabolic Syndrome on in Vitro Fertilization Treatment Outcome
Brief Title: In Vitro Fertilization Outcomes in Metabolic Syndrome
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC-16092013-CTIL
Record Dates: First submitted 2013-10-06; First posted 2013-10-09 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2013-10

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; in vitro fertilization; c reactive protein; over-weight women; ovarian stimulation
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- women with metabolic syndrome: women undergoing ivf treatment who have BMI>25 and meet the criteria for metabolic syndrome
- women without metabolic syndrome: women undergoing ivf treatment who have BMI>25 and who do not meet the criteria for metabolic syndrome

SUMMARY:
The purpose of this study is to examine the effect of metabolic syndrome in over-weight women on IVF treatment outcomes.

DETAILED DESCRIPTION:
This porpuse of the study is to examine the physiology of CRP during the IVF cycle in and to evaluated the effect of CRP in patient with and without metabolic syndrome on IVF outcomes

ELIGIBILITY:
Inclusion Criteria:

* women undergoing ivf treatment

Exclusion Criteria:

* inflammatory disease
* acute conditions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women undergoing ivf treatment in "Meir" medical center in "Kfar-Saba, Israel
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
success or failure of ivf treatment | within 1 year from intiation of ivf treatment
  success or failure of a treatment will be determined by beta-Human chorionic gonadotropin test, number of oocyte retrieved or fertilized and embryos quality.

SECONDARY OUTCOMES:
blood levels of C-reactive protein | within 1 year from initiation of ivf treatment
follicle liquid levels of C-reactive protein | within 1 year from initiation of ivf treatment

CONTACTS AND LOCATIONS:
Overall Officials: Amir Waiser, M.D, Principal Investigator — "Meir", Medical centere
Locations (1):
- Sapir Medical Center, Meir Hospital, Kfar Saba, Israel, Israel

IPD SHARING:
Plan to Share IPD: No